CLINICAL TRIAL: NCT07389382
Title: Effect of Three-Dimensional Educational Material Developed for Pain Mechanisms on Motivation and Knowledge Levels
Brief Title: The Effectiveness of the Three-dimensional Biochemical Activity Model of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Dilek Karaman, Associate Professor, Zonguldak Bulent Ecevit University, Ahmet Erdogan Health Services Vocational School, Health Care Services Program, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 428991-579/24
Record Dates: First submitted 2025-11-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10

CONDITIONS: Pain Management; 3D Printing; Education Nursing
Keywords: Pain Management; 3D Printing; Nursing Students; Education; Motivation to learn
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Students in the intervention group received one hour of training on pain by the same researcher, using a 3D-printed pain biochemical activity model.
  Interventions: Device: 3D printed pain biochemical activity training model
- control group (Other): Students in the control group received one hour of training on pain by the same researcher, using face-to-face instruction and PowerPoint presentations. To avoid interaction between the two laboratories, the control group received training first, followed immediately by the intervention group, who were then transferred to the other laboratory.
  Interventions: Other: PowerPoint Presentations

INTERVENTIONS:
Device: 3D printed pain biochemical activity training model — Computer-generated drawings designed to explain the biochemical mechanism of pain were created using plastic filaments from a 3D printer. Students were divided into small groups of nine using the resulting figures, and the processes of pain mechanisms were explained. At the end of the session, the figures were fixed by applying epoxy resin. After the students poured the epoxy resin onto the models in liquid form, it solidified within six hours, securing the shape as a transparent layer.
  Arms: Intervention group
Other: PowerPoint Presentations — Students in the control group received one hour of training on pain by the same researcher, using face-to-face instruction and PowerPoint presentations. To avoid interaction between the two laboratories, the control group received training first, followed immediately by the intervention group, who were then transferred to the other laboratory.
  Arms: control group

SUMMARY:
Aim: In this study, it was aimed to develop a pain biochemical activity model taken from a three-dimensional printer and fixed by applying epoxy resin and to investigate the effect of this model on nursing students' understanding of the pain mechanism and their motivation to learn.

Methods: The universe of the study consisted of students enrolled in the Biochemistry course at the faculty of nursing of a university in the north of Türkiye during the spring semester of the 2023-2024 academic year. Students were divided into three strata based on their achievement average: high (75 and above), moderate (55-75), and low (54 and below). Forty-five students from each stratum were selected using computer-assisted randomization and assigned to the intervention and control groups. "Student Identification Form", "Pain Mechanism Information Form", "Instructional Material Motivation Scale" and The CONSORT checklist were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Participating voluntarily in the research
* Not having received any previous training in pain
* Being a native Turkish speaker

Exclusion Criteria:

* Being under 18 years old
* Not participating voluntarily in the research
* Having received any previous training in pain
* Not being a native Turkish speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Student Identification Form | This form consisted of six questions and was administered to students one hour prior to the training.
  This form including students' age, gender, high school type, native language, whether they choose a career voluntarily, and whether they have received previous training on pain.
Pain Mechanism Information Form | This form was applied to students 15 minutes before the training began and 5 minutes after the training ended.
  The Pain Mechanism Information Form was developed by the researchers based on literature. The developed questionnaire consists of 14 items, each prepared in a short-answer and fill-in-the-blank format. The scope of the Pain Mechanism Information Form includes: Pain physiology and classification, structure of nociceptors and pain transmission pathways, chemical mediators (Bradykinin, Prostaglandin, Serotonin, CGRP, Substance-P, Histamine), peripheral nerve ending release and mast cell activation, and vascular effects of inflammation (vasodilation, edema).
  Five experts were consulted to ensure the validity of the Pain Mechanism Information Form. Each item was reviewed for its appropriateness and clarity for the intended learning outcomes and content, and necessary revisions were made based on the expert opinions. To ensure reliability, scoring was assessed for short-answer tests, and the questionnaires were scored separately by two raters. The inter-rater reliability coefficient (Cohen'

SECONDARY OUTCOMES:
Instructional Material Motivation Scale | This form was applied to students 30 minutes after the training ended.
  This scale was developed by Tugtekin and Dursun (2022) to measure motivation related to the instructional materials used. It is a one-dimensional, 14-item, 5-point Likert-type self-report scale. High scores on the scale indicate high motivation. The Cronbach's alpha internal consistency coefficient for the measurement tool in this study was determined to be 0.942. Item-total correlation values ranged from 0.629 to 0.820. Permission for use of the scale was obtained from the author via email.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ortiz, M. I., Cuevas-Suarez, C. E., Carino-Cortes, R., de Jesús Navarrete-Hernández, J., & Gonzalez-Montiel, C. A. (2022). Nurses knowledge and attitude regarding pain: A systematic review and meta-analysis. Nurse Education in Practice, 63, 103390.
- [Result] Erickson JM, Brashers V, Owen J, Marks JR, Thomas SM. Effectiveness of an interprofessional workshop on pain management for medical and nursing students. J Interprof Care. 2016 Jul;30(4):466-74. doi: 10.3109/13561820.2016.1159185. Epub 2016 Jun 6. PMID 27268513
- [Result] Murphy-Smith MT, Samawi Z, Abbott P. Teaching Strategies for Nonpharmacological Pain Management to Nursing Students. Pain Manag Nurs. 2024 Oct;25(5):474-479. doi: 10.1016/j.pmn.2024.04.006. Epub 2024 May 6. PMID 38714423
- [Result] Cousins M, Lane-Krebs K, Matthews J, Johnston-Devin C. Student nurses' pain knowledge and attitudes towards pain management over the last 20 years: A systematic review. Nurse Educ Today. 2022 Jan;108:105169. doi: 10.1016/j.nedt.2021.105169. Epub 2021 Oct 9. PMID 34653890
- [Result] Alshehri FA, Levett-Jones T, Pich J. Nursing students' knowledge of and attitudes towards pain management: An integrative review. Nurse Educ Today. 2024 Aug;139:106207. doi: 10.1016/j.nedt.2024.106207. Epub 2024 Apr 10. PMID 38669861
- [Result] Adillon C, Lozano E, Salvat I. Comparison of pain neurophysiology knowledge among health sciences students: a cross-sectional study. BMC Res Notes. 2015 Oct 22;8:592. doi: 10.1186/s13104-015-1585-y. PMID 26493565
- See also: Related Info — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=Murphy-Smith%2C+M.+T.%2C+Samawi%2C+Z.%2C+%26+Abbott%2C+P.+%282024%29.+Teaching+Strategies+for+Nonpharmacological+Pain+Management+to+Nursing+Students.+Pain+Management+Nursing%2C+25%285%29%2C+474-479.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=Alshehri%2C+F.+A.%2C+Levett-Jones%2C+T.%2C+%26+Pich%2C+J.+%282024%29.+Nursing+students%27+knowledge+of+and+attitudes+towards+pain+management%3A+An+integrative+review.+Nurse+Education+Today%2C+106207.&btnG=